CLINICAL TRIAL: NCT03227172
Title: The Accuracy of Magnetic Resonance Imaging in Diagnosing Endodontic Periapical Lesion
Brief Title: Differential Diagnosis Between Granuloma and Radicular Cyst: Effectiveness of Magnetic Resonance Imaging.
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Giuseppe Lizio, research assistant, University of Bologna
Other Study IDs: 15034
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Periapical Diseases
MeSH Terms: conditions — Periapical Diseases | interventions — Apicoectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: apicoectomy — After flap elevation and osteotomy , peri-apical lesion and the root tip were located: after root-end resection using a fissure bur, the resected root tip and the pathological tissue were removed and immediately preserved in 1% formaldehyde solution.

SUMMARY:
The radiolucent periapical jaw lesions of 34 patients, which were surgically enucleated, were investigated by two radiologists using MRI, based on the same six criteria, to categorize the lesions as granulomas or radicular cysts. After apicoectomies, two oral pathologists (blinded to the radiologist's diagnoses) analyzed all specimens by referring to seven specific parameters and diagnosed the specimens as granulomas or radicular cysts. The inter-rater agreements between the radiologists and pathologists in terms of MRI and histological diagnoses, respectively, along with the discriminant power of the adopted criteria and the accuracy of the MRI assessments compared with the histopathologic results, were calculated.

A strong inter-rater reliability was observed between the two radiologists (k-statistic = 0.86, p = 0.0001) and the two pathologists (k-statistic = 0.88, p = 0.0001). Reliability was higher for the radiological (Guttmann's lambda lower bound > 0.6) than histopathological criteria. The accuracy (true positives plus true negatives) of the radiologists was higher than that of the pathologists based on receiver operator characteristic analysis (area under the curve = 0.87 and 0.91, respectively). MRI reliability and accuracy were high and comparable to histopathological reliability, highlighting the usefulness of this non-invasive exam as a pre-treatment diagnostic method for periapical endodontic lesions.

ELIGIBILITY:
Inclusion Criteria:

* patient age ≥ 18 years
* the diameter of the lesion ≥ 5 mm, assessed based on periapical x-ray,
* an acceptable endodontic treatment for the involved tooth.

Exclusion Criteria:

* general medical contraindications for classification of the patient as level III or higher according to the American Society of Anesthesiologists,
* teeth involved in the lesion, the function of which could not be salvaged after enucleation of the lesion and apicoectomy. The radiological exclusion criteria were
* contraindication undergoing magnetic resonance: presence of a pacemaker or any metallic devices that could interfere with the magnetic field;
* severe claustrophobia,
* weight ≥ 130 kg
* intolerance to gadolinium-DTPA as a contrast agent;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 34 patients (17 males and 17 females; mean age 41.9 (range 21-76) years) with periapical endodontic lesions diagnosed by clinical and radiological examination using 2D standard x-rays (periapical and panoramic x-rays) or multislice CT/CBCT in the Oral and Maxillofacial Unit of the University of Bologna between January 2011 and December 2015, and treated with enucleation of the lesion and apicoectomy after a pre-operative MRI exam were retrospectively enrolled in this study. The chart of these patients, that underwent a traditional and standard therapeutic protocol, the radiological imaging and the histopathological data, were analysed after the treatment by a team of two radiologists and two pathologists.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of the resonance magnetic imaging, calculated in comparison with the pathologists' diagnosis with a ROC analysis | 5 years
  To determine the diagnostic accuracy of the radiologists compared with the pathologists (considered the gold standard), receiver operator characteristic (ROC) analysis was performed assuming that the diagnostic test is dichotomous. This method for computing the area under curve (AUC) and its error is in agreement with fitting procedures used for diagnostic tests.

SECONDARY OUTCOMES:
inter-pathologist diagnoses , inter-radiologist diagnoses and internal consistency of the items used for the differential diagnosis by radiologists and pathologists. | 5 years
  To examine inter-rater agreement between the two radiologists and two pathologists, we calculated Cohen's kappa.
  The sensitivity and specificity were determined to assess the ability of MRI to differentially diagnose cysts and granulomas. Sensitivity was calculated as the proportion of true-positive test results (cyst diagnosed consistently by both MRI and biopsy) among the patients with the "disease" (cyst diagnosed by biopsy). Specificity was calculated as the proportion of true-negative results (granuloma diagnosed consistently by both MRI and biopsy) among the "disease-free" subjects (granuloma diagnosed by biopsy) .
  Guttman's lambda coefficient was computed to account for the reliability of the used criteria.

IPD SHARING:
Plan to Share IPD: Undecided